CLINICAL TRIAL: NCT05313607
Title: Effect of Plyometric Exercises on Upper Extremity Function in Children With Unilateral Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amira Mahmoud Abd-elmonem, Amira Abd-elmonem, assist Prof. Physiacl therapy for pediatric department, faculty of physical therapy , Cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: cerebral palsy
Record Dates: First submitted 2022-03-07; First posted 2022-04-06 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Sports Physical Therapy
Keywords: plyometric exercises; Unilateral Cerebral Palsy; cerebral pslay; hand grip strength; upper extremity function; selective motor control
MeSH Terms: interventions — Occupational Therapy; Plyometric Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional group (Experimental): received conventional physical therapy program
  Interventions: Other: Designed physical therapy; Other: Occupational therapy; Other: Conventional Therapy
- plyometric group (Experimental): received a plyometric physical therapy program
  Interventions: Other: Designed physical therapy; Other: Occupational therapy; Other: Plyometric training

INTERVENTIONS:
Other: Designed physical therapy — Attention is given to improve motor function, conducted for 30 minutes
Other: Occupational therapy — included exercises facilitating hand skills, conducted for 30 minutes
Other: Conventional Therapy — aimed to improve the affected upper extremity function, conducted for 30 minutes
  Arms: conventional group
Other: Plyometric training — basically focuses on upper extremity strength training conducted for 30 minutes
  Arms: plyometric group

SUMMARY:
Plyometric training includes muscle contraction that moves rapidly from the eccentric to the concentric phase of movement while using proper biomechanics. It is an effective neuromuscular stimulus that can improve motor functions of children with CP. In plyometric training, muscles exert maximum force in short intervals of time, with the goal of increasing power.

DETAILED DESCRIPTION:
This is a prospective double-masked randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

- spastic hemiplegia

Exclusion Criteria:

- fixed deformities

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Upper extremity function | after 3 successive months
  The quality of upper extremity skill test is used to measure the motor function with maximum score 100% with higher score reflects better performance.
Hand grip strength | after 3 successive months
  The hand held dynamometer was used to assess grip strength and recorded in kilogram.

SECONDARY OUTCOMES:
Selective motor control | after 3 successive months
  Test of arm selective control was used to measure selectivity of upper extremitywith total score for each upper extremity is 16.

CONTACTS AND LOCATIONS:
Overall Officials: walaa A El-nabie, Phd, Study Chair — Cairo university, faculty of physical therapy; Hazem A Ali, Phd, Study Director — Cairo university, faculty of physical therapy
Locations (1):
- Amira Mahmoud Abd-elmonem, Giza, Egypt